CLINICAL TRIAL: NCT00424398
Title: A Single-Center, Double-Masked, Randomized, Placebo-Controlled, Evaluation of the Onset and Duration of Action of Bepotastine Besilate Ophthalmic Solution in Acute Allergic Conjunctivitis
Brief Title: Evaluation of the Onset and Duration of Action of Bepotastine Besilate Ophthalmic Solution in Acute Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISTA-BEPO-CS01
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — bepotastine besilate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Bepreve (Experimental): Bepotastine Besilate Ophthalmic Solution 1.5%
  Interventions: Drug: Bepreve
- Placebo (Placebo Comparator): sterile ophthalmic solution
  Interventions: Drug: Placebo
- Bepotastine Besilate (Experimental): sterile ophthalmic solution 1.0%
  Interventions: Drug: Bepotastine Besilate

INTERVENTIONS:
Drug: Bepreve — sterile ophthalmic solution
  Arms: Bepreve
Drug: Placebo — sterile ophthalmic solution
  Arms: Placebo
Drug: Bepotastine Besilate — sterile ophthalmic solution
  Arms: Bepotastine Besilate

SUMMARY:
The purpose of this study is to evaluate whether bepotastine besilate ophthalmic solution is effective in the treatment of acute allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* At least 10 years of age & either sex, any race
* Willing and able to follow all instructions and attend all study visits
* Positive history of ocular allergies

Exclusion Criteria:

* Have planned surgery during trial period
* Female currently pregnant, planning a pregnancy, or lactating

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-02; Primary Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Williams, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

REFERENCES:
- [Derived] Meier EJ, Torkildsen GL, Gow JA, McNamara TR, Gomes PJ, Williams JI; Bepotastine Besilate Ophthalmic Solutions Study Group. Integrated phase III trials of bepotastine besilate ophthalmic solution 1.5% for ocular itching associated with allergic conjunctivitis. Allergy Asthma Proc. 2012 May-Jun;33(3):265-74. doi: 10.2500/aap.2012.33.3570. PMID 22991696
- [Derived] Torkildsen GL, Williams JI, Gow JA, Gomes PJ, Abelson MB, McNamara TR; Bepotastine Besilate Ophthalmic Solutions Clinical Study Group. Bepotastine besilate ophthalmic solution for the relief of nonocular symptoms provoked by conjunctival allergen challenge. Ann Allergy Asthma Immunol. 2010 Jul;105(1):57-64. doi: 10.1016/j.anai.2010.04.005. PMID 20642205
- [Derived] Abelson MB, Torkildsen GL, Williams JI, Gow JA, Gomes PJ, McNamara TR; Bepotastine Besilate Ophthalmic Solutions Clinical Study Group. Time to onset and duration of action of the antihistamine bepotastine besilate ophthalmic solutions 1.0% and 1.5% in allergic conjunctivitis: a phase III, single-center, prospective, randomized, double-masked, placebo-controlled, conjunctival allergen challenge assessment in adults and children. Clin Ther. 2009 Sep;31(9):1908-21. doi: 10.1016/j.clinthera.2009.09.001. PMID 19843481

RESULTS

PARTICIPANT FLOW:
Groups:
- Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5%; Placebo; Bepotastine Besilate Ophthalmic Solution 1.0%: 1 drop, both eyes at 3 different time points post-CAC within 3 different time points post-dose, for a total of 9 separate time points
Period: Overall Study
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Started | 35 | 36 | 36
Completed | 32 | 35 | 36
Not Completed | 3 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Subject met exclusion criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0% | Total
Number analyzed (Participants) | 35 | 36 | 36 | 107
Age, Customized [Number; unit: participants]
  <18 years | 2 | 2 | 3 | 7
  >=18 years | 33 | 34 | 33 | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 44.3 (16.0) | 40.9 (11.4) | 39.9 (15.2) | 41.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 14 | 49
  Male | 17 | 19 | 22 | 58

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular Itching score: 0=None; 0.5=Intermittent tickle sensation possibly localized in the corner of the eye; 1.0=Intermittent tickle sensation involving more than the corner of the eye; 1.5=Intermittent all-over tickling sensation; 2.0=Mild continuous itch (can be localized) without desire to rub; 2.5=Moderate, diffuse continuous itch with desire to rub; 3.0=Severe itch with desire to rub; 3.5=Severe itch improved with minimal rubbing; 4.0=Incapacitating itch with irresistible urge to rub
Time Frame: 15 minutes, 8 hours & 16 hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 3 Minutes post CAC | 0.5 (0.8) | 1.9 (0.8) | 0.6 (0.7)
  15 Minutes post-dose: 5 Minutes post CAC | 0.8 (0.9) | 2.1 (0.8) | 0.7 (0.8)
  15 Minutes post-dose: 7 Minutes post CAC | 0.7 (0.9) | 2.0 (0.7) | 0.7 (0.8)
  8 Hours post-dose: 3 Minutes post CAC | 0.8 (0.9) | 2.0 (0.7) | 1.2 (0.8)
  8 Hours post-dose: 5 Minutes post CAC | 0.9 (1.0) | 2.3 (0.7) | 1.3 (0.8)
  8 Hours post-dose: 7 Minutes post CAC | 0.9 (1.0) | 2.2 (0.8) | 1.3 (0.8)
  16 Hours post-dose: 3 Minutes post CAC | 1.3 (1.0) | 2.1 (0.9) | 1.4 (0.7)
  16 Hours post-dose: 5 Minutes post CAC | 1.5 (1.1) | 2.4 (0.8) | 1.6 (0.9)
  16 Hours post-dose: 7 Minutes post CAC | 1.5 (1.0) | 2.3 (0.8) | 1.4 (1.0)

2. Primary Outcome: Conjunctival Redness
Description: Conjunctival Redness score: 0=None; 1.0=Mild-Slightly dilated blood vessels; color of vessels typically pink; 2.0=Moderate-More apparent dilation of blood vessels; vessel color more intense (redder); 3.0=Severe-Numerous, obvious dilated blood vessels; absence of chemosis color is deep red, presence of chemosis may be less red or pink; 4.0=Extremely Severe-Large, numerous dilated blood vessels characterized by severe deep red color regardless of chemosis grade
Time Frame: 15 minutes, 8 hours & 16 hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 1.4 (0.8) | 1.9 (0.6) | 1.1 (0.7)
  15 Minutes post-dose: 15 Minutes post CAC | 1.7 (0.8) | 2.1 (0.6) | 1.5 (0.7)
  15 Minutes post-dose: 20 Minutes post CAC | 1.6 (0.8) | 2.0 (0.6) | 1.4 (0.7)
  8 Hours post-dose: 7 Minutes post CAC | 1.3 (0.7) | 1.7 (0.7) | 1.3 (0.6)
  8 Hours post-dose: 15 Minutes post CAC | 1.5 (0.8) | 1.9 (0.6) | 1.6 (0.6)
  8 Hours post-dose: 20 Minutes post CAC | 1.6 (0.8) | 1.9 (0.7) | 1.6 (0.7)
  16 Hours post-dose: 7 Minutes post CAC | 1.7 (0.5) | 1.8 (0.6) | 1.4 (0.6)
  16 Hours post-dose: 15 Minutes post CAC | 1.9 (0.6) | 1.8 (0.6) | 1.5 (0.7)
  16 Hours post-dose: 20 minutes post CAC | 1.8 (0.6) | 1.7 (0.6) | 1.5 (0.7)

3. Secondary Outcome: Ciliary Redness
Description: Ciliary Redness score: 0=None; 1.0=Mild-Slightly dilated blood vessels; color of vessels typically pink; 2.0=Moderate-More apparent dilation of blood vessels; vessel color more intense (redder); 3.0=Severe-Numerous, obvious dilated blood vessels; absence of chemosis color is deep red, presence of chemosis may be less red or pink; 4.0=Extremely Severe-Large, numerous dilated blood vessels characterized by severe deep red color regardless of chemosis grade
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minute post CAC | 1.2 (0.9) | 1.7 (0.6) | 0.9 (0.7)
  15 Minutes post-dose: 15 Minute post CAC | 1.5 (0.9) | 1.9 (0.6) | 1.3 (0.8)
  15 Minutes post-dose: 20 Minute post CAC | 1.6 (0.8) | 1.8 (0.7) | 1.3 (0.8)
  8 Hours post-dose: 7 Minute post CAC | 1.2 (0.8) | 1.5 (0.7) | 1.2 (0.7)
  8 Hours post-dose: 15 Minute post CAC | 1.5 (0.9) | 1.7 (0.7) | 1.5 (0.7)
  8 Hours post-dose: 20 Minute post CAC | 1.4 (0.9) | 1.7 (0.7) | 1.4 (0.8)
  16 Hours post-dose: 7 Minute post CAC | 1.6 (0.7) | 1.7 (0.6) | 1.3 (0.7)
  16 Hours post-dose: 15 Minute post CAC | 1.9 (0.7) | 1.9 (0.6) | 1.5 (0.7)
  16 Hours post-dose: 20 Minute post CAC | 1.7 (0.7) | 1.8 (0.7) | 1.4 (0.8)

4. Secondary Outcome: Episcleral Redness
Description: Episcleral Redness score: 0=None; 1.0=Mild-Slightly dilated blood vessels; color of vessels typically pink; 2.0=Moderate-More apparent dilation of blood vessels; vessel color more intense (redder); 3.0=Severe-Numerous, obvious dilated blood vessels; absence of chemosis color is deep red, presence of chemosis may be less red or pink; 4.0=Extremely Severe-Large, numerous dilated blood vessels characterized by severe deep red color regardless of chemosis grade
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 1.3 (0.8) | 1.9 (0.6) | 1.1 (0.7)
  15 Minutes post-dose: 15 Minutes post CAC | 1.6 (0.8) | 2.1 (0.6) | 1.5 (0.7)
  15 Minutes post-dose: 20 Minutes post CAC | 1.6 (0.8) | 2.0 (0.7) | 1.4 (0.7)
  8 Hours post-dose: 7 Minutes post CAC | 1.4 (0.7) | 1.7 (0.7) | 1.4 (0.6)
  8 Hours post-dose: 15 Minutes post CAC | 1.6 (0.8) | 1.9 (0.6) | 1.7 (0.6)
  8 Hours post-dose: 20 Minutes post CAC | 1.6 (0.8) | 1.9 (0.7) | 1.6 (0.7)
  16 Hours post-dose: 7 Minutes post CAC | 1.8 (0.5) | 2.0 (0.5) | 1.4 (0.7)
  16 Hours post-dose: 15 Minutes post CAC | 1.9 (0.7) | 2.0 (0.5) | 1.6 (0.7)
  16 Hours post-cose: 20 Minutes post CAC | 1.9 (0.6) | 1.9 (0.6) | 1.5 (0.8)

5. Secondary Outcome: Chemosis
Description: Chemosis score: 0 = None; 1.0 = Mild-Detectable only by slit lamp beam; definite separation of conjunctiva from sclera; 2.0 = Moderate-Visible in normal room light; more diffuse edema; 3.0 = Severe-Conjunctival billowing at the limbus; very diffuse and noticeable; 4.0 = Extremely Severe-Overall ballooning of conjunctiva
Time Frame: 15 Minutes, 8 Hours & s6 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.4 (0.3) | 0.7 (0.5) | 0.4 (0.3)
  15 Minutes post-dose: 15 Minutes post CAC | 0.6 (0.5) | 0.9 (0.6) | 0.5 (0.3)
  15 Minutes post-dose: 20 Minutes post CAC | 0.5 (0.3) | 0.8 (0.6) | 0.5 (0.3)
  8 Hours post-dose: 7 Minutes post CAC | 0.5 (0.5) | 0.7 (0.5) | 0.5 (0.4)
  8 Hours post-dose: 15 Minutes post CAC | 0.8 (0.7) | 0.9 (0.6) | 0.7 (0.4)
  8 Hours psot-dose: 20 Minutes post CAC | 0.8 (0.7) | 0.9 (0.6) | 0.8 (0.4)
  16 Hours post-dose: 7 Minutes post CAC | 0.7 (0.5) | 0.9 (0.4) | 0.6 (0.4)
  16 Hours post-dose: 15 Minutes post CAC | 0.9 (0.5) | 1.1 (0.5) | 0.8 (0.4)
  16 Hours post-dose: 20 Minutes post CAC | 0.9 (0.6) | 1.1 (0.6) | 0.8 (0.5)

6. Secondary Outcome: Rhinorrhea (Runny Nose)
Description: Rhinorrhea score: 0 = None; 1.0 = Mild-Sensation of nasal mucus flowing down nasal passage; no discharge present; 2.0 = Moderate-May be associated with post-nasal drip; nasal mucus flow more pronounced; will need to blow nose soon; 3.0 = Moderate/Severe-Nasal mucus discharge requiring occasional wiping with Kleenex; 4.0 = Severe-Uncontrolled nasal discharge; requiring frequent wiping and blowing nose
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.4 (0.8) | 0.9 (1.0) | 0.1 (0.3)
  15 Minutes post-dose: 15 Minutes post CAC | 0.5 (0.9) | 1.1 (1.0) | 0.2 (0.6)
  15 Minutes post-dose: 20 Minutes post CAC | 0.4 (0.8) | 0.9 (1.1) | 0.3 (0.6)
  8 Hours post-dose: 7 Minutes post CAC | 0.2 (0.5) | 0.9 (1.0) | 0.3 (0.7)
  8 Hours post-dose: 15 Minutes post CAC | 0.3 (0.6) | 1.5 (1.2) | 0.5 (0.8)
  8 Hours post-dose: 20 Minutes post CAC | 0.3 (0.6) | 1.3 (1.3) | 0.4 (0.7)
  16 Hours post-dose: 7 Minutes post CAC | 0.4 (0.7) | 1.0 (1.0) | 0.4 (0.8)
  16 Hours post-dose: 15 Minutes post CAC | 0.6 (0.8) | 1.4 (1.1) | 0.8 (0.9)
  16 Hours post-dose: 20 Minutes post CAC | 0.7 (0.9) | 1.2 (1.2) | 0.8 (1.0)

7. Secondary Outcome: Nasal Pruritus (Itchy Nose)
Description: Nasal Pruritus score: 0 = None; 1.0 = Mild-An intermittent tickle sensation; 2.0 = Moderate-A mild continuous itch; 3.0 = Moderate/Severe-A severe itch with desire to rub; 4.0 = Severe-Incapacitating itch with an irresistible urge to rub
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.3 (0.7) | 0.7 (0.8) | 0.1 (0.3)
  15 Minutes post-dose: 15 Minutes post CAC | 0.2 (0.6) | 0.9 (0.8) | 0.2 (0.5)
  15 Minutes post-dose: 20 Minutes post CAC | 0.2 (0.6) | 0.6 (0.8) | 0.3 (0.6)
  8 Hours post-dose: 7 Minutes post CAC | 0.1 (0.4) | 0.6 (0.9) | 0.3 (0.7)
  8 Hours post-dose: 15 Minutes post CAC | 0.2 (0.5) | 0.9 (1.1) | 0.3 (0.6)
  8 Hours post-dose: 20 Minutes post CAC | 0.3 (0.6) | 0.8 (1.1) | 0.3 (0.6)
  16 Hours post-dose: 7 Minutes post CAC | 0.5 (0.7) | 0.8 (1.0) | 0.3 (0.6)
  16 Hours post-dose: 15 Minutes post CAC | 0.5 (0.9) | 0.9 (1.1) | 0.4 (0.6)
  16 Hours post-dose: 20 Minutes post CAC | 0.5 (0.9) | 0.8 (1.1) | 0.4 (0.7)

8. Secondary Outcome: Ear or Palate Pruritus (Itchy Ear or Palate)
Description: Ear or Palate Pruritus score: 0 = None; 1.0 = Mild-An intermittent tickle sensation; 2.0 = Moderate-A mild continuous itch; 3.0 = Moderate/Severe-A severe itch with desire to rub; 4.0 = Severe-Incapacitating itch with an irresistible urge to rub
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.3 (0.7) | 0.6 (0.9) | 0.1 (0.2)
  15 Minutes post-dose: 15 Minutes post CAC | 0.6 (0.9) | 0.9 (1.0) | 0.2 (0.5)
  15 Minutes post-dose: 20 Minutes post CAC | 0.6 (0.9) | 0.9 (1.0) | 0.3 (0.6)
  8 Hours post-dose: 7 Minutes post CAC | 0.2 (0.5) | 0.6 (0.9) | 0.4 (0.8)
  8 Hours post-dose: 15 Minutes post CAC | 0.4 (0.9) | 1.2 (1.2) | 0.4 (0.8)
  8 Hours post-dose: 20 Minutes post CAC | 0.5 (0.8) | 0.9 (1.1) | 0.5 (0.9)
  16 Hours post-dose: 7 Minutes post CAC | 0.5 (0.7) | 0.6 (0.9) | 0.3 (0.8)
  16 Hours post-dose: 15 Minutes post CAC | 0.8 (1.0) | 1.0 (1.2) | 0.8 (1.2)
  16 Hours post-dose: 20 Minutes post CAC | 0.8 (1.0) | 0.9 (1.2) | 0.8 (1.1)

9. Secondary Outcome: Nasal Congestion
Description: Nasal Congestion score: 0 = None-Breathes freely; 1.0 = Mild-Breathes with difficulty; 2.0 = Moderate-One nostril partially blocked; 3.0 = Moderate/Severe-Both nostrils partially blocked or one nostril completely blocked and the other nostril partially blocked; 4.0 = Severe-Both nostrils completely blocked
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.5 (1.0) | 0.9 (1.0) | 0.2 (0.4)
  15 Minutes post-dose: 15 Minutes post CAC | 0.4 (0.9) | 1.1 (1.2) | 0.3 (0.6)
  15 Minutes post-dose: 20 Minutes post CAC | 0.4 (0.9) | 1.2 (1.1) | 0.3 (0.5)
  8 Hours post-dose: 7 Minutes post CAC | 0.2 (0.5) | 0.9 (1.0) | 0.3 (0.6)
  8 Hours post-dose: 15 Minutes post CAC | 0.4 (0.8) | 1.2 (1.2) | 0.4 (0.7)
  8 Hours post-dose: 20 Minutes post CAC | 0.4 (0.8) | 1.1 (1.2) | 0.4 (0.7)
  16 Hours post-dose: 7 Minutes post CAC | 0.4 (0.7) | 1.0 (1.0) | 0.4 (0.8)
  16 Hours post-dose: 15 Minutes post CAC | 0.7 (1.0) | 1.3 (1.1) | 0.8 (1.0)
  16 Hours post-dose: 20 Minutes post CAC | 0.7 (1.0) | 1.2 (1.2) | 0.8 (1.0)

10. Secondary Outcome: Tearing
Description: Percent of Eyes with Tearing. Scored as absent or present
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Number; unit: Percent of Eyes with Tearing Present
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Percent of Eyes with Tearing Present
  15 Minutes post-dose: 7 Minutes post CAC | 14.3 | 43.1 | 6.9
  15 Minutes post-dose: 15 Minutes post CAC | 17.1 | 34.7 | 9.7
  15 Minutes post-dose: 20 Minutes post CAC | 17.1 | 38.9 | 11.1
  8 Hours post-dose: 7 Minutes post CAC | 12.9 | 50.0 | 13.9
  8 Hours post-dose: 15 Minutes post CAC | 14.3 | 56.9 | 16.7
  8 Hours post-dose: 20 Minutes post CAC | 12.9 | 40.3 | 15.3
  16 Hours post-dose: 7 Minutes post CAC | 11.4 | 43.1 | 23.6
  16 Hours post-dose: 15 Minutes post CAC | 15.7 | 44.4 | 19.4
  16 Hours post-dose: 20 Minutes post CAC | 15.7 | 34.7 | 23.6

11. Secondary Outcome: Ocular Mucus Discharge
Description: Percent of Eyes with Ocular Mucus Discharge. Scored as absent or present
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Number; unit: Percent of Eyes with OMD Present
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Percent of Eyes with OMD Present
  15 Minutes post-dose: 7 Minutes post CAC | 0.0 | 1.4 | 0.0
  15 Minutes post-dose: 15 Minutes post CAC | 2.9 | 0.0 | 0.0
  15 Minutes post-dose: 20 Minutes post CAC | 2.9 | 0.0 | 0.0
  8 Hours post-dose: 7 Minutes post CAC | 0.0 | 1.4 | 1.4
  8 Hours post-dose: 15 Minutes post CAC | 0.0 | 2.8 | 1.4
  8 Hours post-dose: 20 Minutes post CAC | 0.0 | 2.8 | 0.0
  16 Hours post-dose: 7 Minutes post CAC | 0.0 | 2.8 | 0.0
  16 Hours post-dose: 15 Minutes post CAC | 0.0 | 5.6 | 0.0
  16 Hours post-dose: 20 Minutes post CAC | 0.0 | 5.6 | 0.0

12. Secondary Outcome: Eyelid Swelling
Description: Eyelid Swelling score: 0 = None; 1.0 = Mild-Detectable swelling of lower and/or upper lid; 2.0 = Moderate-Definite swelling of lower and/or upper lid; 3.0 = Severe-Swelling of lower and/or upper lid to the point that there is a decrease in the space between your upper and lower lids
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.3 (0.5) | 0.7 (0.7) | 0.2 (0.5)
  15 Minutes post-dose: 15 Minutes post CAC | 0.3 (0.5) | 0.8 (0.7) | 0.2 (0.6)
  15 Minutes post-dose: 20 Minutes post CAC | 0.3 (0.5) | 0.9 (0.7) | 0.3 (0.6)
  8 Hours post-dose: 7 Minutes post CAC | 0.4 (0.7) | 0.7 (0.7) | 0.3 (0.5)
  8 Hours post-dose: 15 Minutes post CAC | 0.5 (0.8) | 0.9 (0.9) | 0.4 (0.6)
  8 Hours post-dose: 20 Minutes post CAC | 0.5 (0.7) | 0.9 (0.9) | 0.4 (0.6)
  16 Hours post-dose: 7 Minutes post CAC | 0.5 (0.6) | 0.7 (0.7) | 0.3 (0.5)
  16 Hours post-dose: 15 Minutes post CAC | 0.5 (0.7) | 0.9 (0.9) | 0.4 (0.6)
  16 Hours post-dose: 20 Minutes post CAC | 0.5 (0.7) | 0.8 (0.8) | 0.5 (0.6)

13. Secondary Outcome: Total Nasal Symptom
Description: Total Nasal Symptom score (Composite of Rhinorrhea, Nasal Pruritus, Ear or Palate Pruritus, and Nasal Congestion): 0 = None; 1.0 = Mild; 2.0 = Moderate; 3.0 = Moderate/Severe; 4.0 = Severe
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 35 | 36 | 36
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 1.3 (2.2) | 3.2 (3.1) | 0.4 (0.8)
  15 Minutes post-dose: 15 Minutes post CAC | 1.7 (2.2) | 4.0 (3.4) | 0.9 (1.5)
  15 Minutes post-dose: 20 Minutes post CAC | 1.6 (2.2) | 3.6 (3.2) | 1.0 (1.6)
  8 Hours post-dose: 7 Minutes post CAC | 0.7 (1.6) | 2.9 (3.1) | 1.3 (2.4)
  8 Hours post-dose: 15 Minutes post CAC | 1.3 (2.2) | 4.8 (4.0) | 1.6 (2.5)
  8 Hours post-dose: 20 Minutes post CAC | 1.5 (2.4) | 4.0 (4.0) | 1.5 (2.4)
  16 Hours post-dose: 7 Minutes post CAC | 1.8 (2.0) | 3.4 (3.2) | 1.3 (2.6)
  16 Hours post-dose: 15 Minutes post CAC | 2.5 (2.9) | 4.5 (4.0) | 2.7 (3.1)
  16 Hours post-dose: 20 Minutes post CAC | 2.6 (3.1) | 4.0 (4.3) | 2.8 (3.3)

ADVERSE EVENTS:
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 4/35 | 2/36 | 8/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% (N=35) | Placebo (N=36) | Bepotastine Besilate Ophthalmic Solution 1.0% (N=36)
Mild Taste (Nervous system disorders) | 3 | 0 | 6
Eye Irritation (Eye disorders) | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement is between contract research organization and third parties on behalf of ISTA Pharmaceuticals, Inc.